CLINICAL TRIAL: NCT00180596
Title: Pacing for Cardiomyopathies, a European Study- A Therapy Acceptance Study
Brief Title: PACMAN - PAcing for CardioMyopathies, a EuropeAN Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PACMAN-1099
Record Dates: First submitted 2005-09-15; First posted 2005-09-16 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2005-06

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

INTERVENTIONS:
Device: Contak heart failure devices

SUMMARY:
The purpose of this study was to evaluate the benefit of biventricular pacing in patients with heart failure who were receiving optimal pharmacological therapy, and who were either with or without an ICD indication

DETAILED DESCRIPTION:
Heart Failure is a syndrome that affects millions of patients in Europe with over half a million new cases reported annually. Drug therapy had been the conventional treatment of choice until the emergence of cardiac resynchronization therapy (CRT) where biventricular pacing can be delivered to the heart through a pacemaker or implantable cardioverter defibrillator. This study was designed to assess the effect of CRT on patients optimized on conventional heart failure medication including diuretics, beta blockers and ACE inhibitors. The effect of CRT was evaluated by comparison of 6 minute walk performance, Quality of Life and NHYA class after 6 months with CRT therapy either programmed ON or OFF. In addition, evaluation of the incidence of adverse events (predefined as ventricular arrhythmias, hospitalizations, drop-outs, complications and patient deaths) was done between groups at 6 months. Patients were all programmed ON after 6 months and data was collected for an additional 6 months.

ELIGIBILITY:
Inclusion Criteria:

- NYHA Class III and IV with EF < 35%; Optimal individual drug therapy in 2 weeks prior to enrollment including ACE inhibitors; beta blockers and diuretics unless not tolerated

Exclusion Criteria:

* Reduced life expectancy of < 6 months or candidate for heart transplant within 6 months; chronic/recurrent atrial fibrillation/flutter

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262
Dates: Start 2000-01; Study Completion 2005-09

PRIMARY OUTCOMES:
Improvement in functional capacity as measured by a six-minute walk test at 6 months

SECONDARY OUTCOMES:
Improvement in Quality of Life at 6 months; Improvement in NHYA classification at 6 months; incidence of adverse events at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: P HANRATH, MD, Principal Investigator — Medizinische Klinik I, University RWTH Aachen, Pauwelsstr. 30, 52057 Aachen, Germany
Locations (2):
- Guidant Corporation, , , Belgium, Diegem, Belgium
- Medizinische Klinik I, University RWTH Aachen, Aachen, Germany